CLINICAL TRIAL: NCT02891954
Title: Pharmacogenomics to Predict Responses to SGLT2 Inhibitors
Brief Title: Genetics of Response to Canagliflozin
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Simeon I. Taylor, Professor of Medicine, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HP-00069977; R01DK118942 (NIH)
Record Dates: First submitted 2016-08-30; First posted 2016-09-08 (Estimated); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Glucosuria; SGLT2 inhibitors; Canagliflozin; FGF23; Parathyroid hormone; 1,25-Dihydroxyvitamin D; Glucagon; Ketone bodies; Uric acid; Pharmacogenomics
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Glycosuria | interventions — Canagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm (Experimental): Healthy volunteers will receive canagliflozin to assess pharmacodynamic responses to drug.
  Interventions: Drug: Canagliflozin

INTERVENTIONS:
Drug: Canagliflozin — Healthy volunteers will receive canagliflozin (300 mg per day) in the morning for five days.
  Other Names: Invokana (brand name for canagliflozin)

SUMMARY:
Five daily doses of canagliflozin (300 mg) will be administered to healthy volunteers. Pharmacodynamic responses to canagliflozin will be assessed both at 2 days and 6 days after administration of the first dose of canagliflozin. A genome-wide association study (GWAS) will be conducted to search for genetic variants that are associated with each of the pharmacodynamic responses to canagliflozin.

DETAILED DESCRIPTION:
After obtaining informed consent, healthy Amish research subjects will be screened for eligibility. Immediately after obtaining blood samples for baseline clinical chemistry tests wills, patients will initiate 5 days of canagliflozin (300 mg) treatment. Fasting blood samples will be obtained to assess pharmacodynamic responses at both 48 hours and 120 hours after initiating canagliflozin. The principal pharmacodynamic responses will include 24 hour urinary excretion of glucose, serum chemistries (phosphorus, FGF23, 1,25-dihydroxyvitamin D, parathyroid hormone (PTH), glucagon, beta-hydroxybutyrate, acetoacetate, procollagen type I N-terminal peptide (P1NP), and beta-CTX). Research subjects will undergo genotyping, and a genome-wide association study will be conducted to search for genetic variants that are associated with pharmacodynamic responses to canagliflozin.

ELIGIBILITY:
Inclusion Criteria:

* Of Amish descent
* Age 18 or older
* BMI: 18-40 kg/m2

Exclusion Criteria:

* Known allergy to canagliflozin
* History of diabetes, random glucose greater than 200 mg/dL, or HbA1c greater than or equal to 6.5%
* Currently taking diuretics, antihypertensive medication uric acid lowering medications, or other medication that the investigator judges will make interpretation of the results difficult
* Significant debilitating chronic cardiac, hepatic, pulmonary, or renal disease or other diseases that the investigator judges will make interpretation of the results difficult or increase the risk of participation
* Seizure disorder
* Unwilling to go off of vitamin supplements and over the counter medication (except for acetaminophen) for at least two weeks prior to the first home visit and agree to avoid these medications for the duration of the study.
* Positive urine human chorionic gonadotropin test or known pregnancy within 3 months of the start of the study
* Estimated glomerular filtration rate less than 60 mL/min
* Currently breast feeding or breast feeding within 3 month of the start of the study
* Liver function tests greater than 2 times the upper limit of normal
* Hematocrit less than 35%
* Abnormal thyroid hormone stimulating hormone

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2016-09 (Actual); Primary Completion 2023-09-25 (Actual); Study Completion 2026-12-25 (Estimated)

PRIMARY OUTCOMES:
Urinary glucose excretion (during the time interval 24-48 hours after first administration of canagliflozin) | 24-48 hours
  Urine collection will be initiated 24 hours after initiation of canagliflozin treatment, and continued for an additional 24 hours.

SECONDARY OUTCOMES:
Bone-related biomarkers | 48 hrs
  Serum phosphorus, FGF23, 1,25-dihydroxyvitamin D, PTH, P1NP, and beta-CTX
Bone-related biomarkers | 120 hrs
  Serum phosphorus, FGF23, 1,25-dihydroxyvitamin D, PTH, P1NP, and beta-CTX
Ketosis-related biomarkers | 48 hrs
  glucagon, acetoacetate, beta-hydroxybutyrate
Ketosis-related biomarkers | 120 hurs
  glucagon, acetoacetate, beta-hydroxybutyrate
Serum uric acid | 48 hrs
  Change in serum uric acid at 48 hours
Serum uric acid | 120 hrs
  Change in serum uric acid at 120 hours

CONTACTS AND LOCATIONS:
Overall Officials: Simeon I Taylor, MD, PhD, Principal Investigator — Unversity of Maryland School of Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Taylor SI, Blau JE, Rother KI. Possible adverse effects of SGLT2 inhibitors on bone. Lancet Diabetes Endocrinol. 2015 Jan;3(1):8-10. doi: 10.1016/S2213-8587(14)70227-X. Epub 2014 Dec 16. No abstract available. PMID 25523498
- [Background] Taylor SI, Blau JE, Rother KI. SGLT2 Inhibitors May Predispose to Ketoacidosis. J Clin Endocrinol Metab. 2015 Aug;100(8):2849-52. doi: 10.1210/jc.2015-1884. Epub 2015 Jun 18. PMID 26086329
- [Background] Blau JE, Bauman V, Conway EM, Piaggi P, Walter MF, Wright EC, Bernstein S, Courville AB, Collins MT, Rother KI, Taylor SI. Canagliflozin triggers the FGF23/1,25-dihydroxyvitamin D/PTH axis in healthy volunteers in a randomized crossover study. JCI Insight. 2018 Apr 19;3(8):e99123. doi: 10.1172/jci.insight.99123. eCollection 2018 Apr 19. PMID 29669938
- [Background] Blau JE, Taylor SI. Adverse effects of SGLT2 inhibitors on bone health. Nat Rev Nephrol. 2018 Aug;14(8):473-474. doi: 10.1038/s41581-018-0028-0. PMID 29875481
- [Background] Beitelshees AL, Leslie BR, Taylor SI. Sodium-Glucose Cotransporter 2 Inhibitors: A Case Study in Translational Research. Diabetes. 2019 Jun;68(6):1109-1120. doi: 10.2337/dbi18-0006. PMID 31109940
- [Result] Shahidzadeh Yazdi Z, Streeten EA, Whitlatch HB, Montasser ME, Beitelshees AL, Taylor SI. Vitamin D Deficiency Increases Vulnerability to Canagliflozin-induced Adverse Effects on 1,25-Dihydroxyvitamin D and PTH. J Clin Endocrinol Metab. 2024 Jan 18;109(2):e646-e656. doi: 10.1210/clinem/dgad554. PMID 37738423
- [Result] Shahidzadeh Yazdi Z, Streeten EA, Whitlatch HB, Montasser ME, Beitelshees AL, Taylor SI. Critical Role for 24-Hydroxylation in Homeostatic Regulation of Vitamin D Metabolism. J Clin Endocrinol Metab. 2025 Jan 21;110(2):e443-e455. doi: 10.1210/clinem/dgae156. PMID 38481375
- [Result] Shahidzadeh Yazdi Z, Streeten EA, Whitlatch HB, Bargal SA, Beitelshees AL, Taylor SI. Value of Vitamin D Metabolite Ratios in 3 Patients as Diagnostic Criteria to Assess Vitamin D Status. JCEM Case Rep. 2024 Jun 28;2(7):luae095. doi: 10.1210/jcemcr/luae095. eCollection 2024 Jul. PMID 38947416
- [Derived] Taylor SI, Cherng HR, Shahidzadeh Yazdi Z, Montasser ME, Whitlatch HB, Mitchell BD, Shuldiner AR, Streeten EA, Beitelshees AL. Pharmacogenetics of sodium-glucose co-transporter-2 inhibitors: Validation of a sex-agnostic pharmacodynamic biomarker. Diabetes Obes Metab. 2023 Dec;25(12):3512-3520. doi: 10.1111/dom.15246. Epub 2023 Aug 22. PMID 37608471